CLINICAL TRIAL: NCT04625153
Title: RC18, a Recombinant Human B Lymphocyte Stimulator Receptor:Immunoglobulin G( IgG ) Fc Fusion Protein for Injection in Patients With Relapsing Remitting Multiple Sclerosis：a Phase II Trial
Brief Title: RC18 in Patients With Relapsing Remitting Multiple Sclerosis：a Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18C013
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — RC-18; telitacicept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC18 160mg (Experimental): RC18 160mg is injected subcutaneously once a week for 48 times.
  Interventions: Biological: RC18 160mg
- RC18 240mg (Experimental): RC18 240mg is injected subcutaneously once a week for 48 times.
  Interventions: Biological: RC18 240mg

INTERVENTIONS:
Biological: RC18 160mg — RC18 160mg is injected subcutaneously once a week for 48 times.
  Other Names: telitacicept
  Arms: RC18 160mg
Biological: RC18 240mg — RC18 240mg is injected subcutaneously once a week for 48 times.
  Other Names: telitacicept
  Arms: RC18 240mg

SUMMARY:
To observe the safety and effectivity of a Recombinant Human B Lymphocyte Stimulator Receptor : Immunoglobulin G( IgG ) Fc Fusion Protein for injection (RC18) in patients with relapsing remitting multiple sclerosis, analyze the dose-response relationship and provide a dose basis for follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing remitting multiple sclerosis meet the diagnostic criteria of McDonald 2017.
* 18-55 years old, male or female
* At least 1 recurrence was recorded within 1 year prior to randomization, or at least 2 recurrences within 2 years (the first clinical episode of MS was recorded as a recurrence), or active gadolinium enhanced lesions in the brain within 1 year prior to screening.
* Neurological symptoms were stable for ≥30 days before screening and before baseline
* EDSS score ≤ 5.5
* Informed consent signed voluntarily

Exclusion Criteria:

* Patients who were unable to undergo magnetic resonance imaging or who were allergic to gadolinium contrast agents during the trial
* In addition to multiple sclerosis, patients with chronic active immune system diseases or who are stable but require immunotherapy (glucocorticoids and/or immunosuppressants) (e.g., rheumatoid arthritis, scleroderma, Sjogren's syndrome, Crohn's disease, ulcerative colitis), Or patients with known immunodeficiency syndromes (AIDS, genetic immunodeficiency, and drug-induced immunodeficiency); Patients who received glucocorticoid maintenance therapy before randomization could participate in the trial after discontinuing the drug.
* Patients who were AQP4 antibody positive and/or MOG antibody positive within 1 year prior to randomization
* Patients who have received the following treatment:

  1. Interferon, pegylated interferon, glatirex acetate, and dimethyl fumarate were used within 4 weeks prior to randomization.
  2. Use of Fingomod, intravenous immunoglobulin, or plasmapheresis within 12 weeks prior to randomization.
  3. Alemtuzumab, Daclizumab, Ocrelizumab were administered within 24 weeks prior to randomization.
  4. Azathioprine (AZA, half-life t1/2=6hrs), Mycophenolate Mofetil (t1/2=16hrs), Leflunomide (LEF, LEflunomide) were used before randomization. t1/2=15 days), Tacrolimus (t1/2=43 hrs), Teriflunomide (t1/2=18 days), Cyclosporin (CsA) Patients with immunosuppressants such as t1/2=27 hrs), Methotrexate (MTX, t1/2=14hrs), Cyclophosphamide (CTX, t1/2=6hrs), in addition to leflunomide and teriflunomide, The discontinuation interval was more than 5 times the half-life. Leflunomide and Teriflunomide need to be eluted with coletenide, which can be discontinued and the following measures taken: Coletenide 8 g 3 times daily for 11 days, if the 8 g dose is not tolerated, can be changed to 4 g orally for the same time and frequency as before.
  5. Use of clatribine or mitoxantrone within 1 year prior to randomization.
  6. Received lymphoid irradiation and bone marrow transplantation before randomization.
* Patients were participated in any clinical trial 28 days before randomization or within 5 times half-life of study drug participating in clinical trial (whichever is longer).
* Patients with any persistent or chronic active infection or serious infection history in the screening period, such as shingles; active tuberculosis (patients with latent tuberculosis can participate in the test if they are given isoniazid and / or rifampin at the same time); HIV infection; syphilis antibody positive; HCV antibody positive; HBsAg positive; HBsAg negative but HBcAb positive, the HBV-DNA quantitative test is needed. If the HBV-DNA is positive, the patient should be excluded. If the HBV-DNA is negative, the patient can not be excluded.
* The results of abnormal laboratory tests to be excluded include but are not limited to: Leukocyte count < 3 × 10~9 / L; neutrophil < 1.5 × 10~9 / L; hemoglobin < 85g / L; platelet count < 80 × 10~9 / L; serum creatinine > 1.5 × ULN, accompanied by creatinine clearance < 50ml / min (measured value, or calculated by Cockcroft Gault formula); total bilirubin > 1.5 × ULN; ALT > 3 × ULN; AST > 3 × ULN; alkaline phosphatase > 2 × ULN; IgG < lower limit of normal value; IgM < lower limit of normal value;
* Cancer patients
* Pregnant women, lactating women and patients with family planning during the trial
* Patients with other mental disorders
* Patients who experienced any of the following events within 12 weeks before randomization: myocardial infarction, unstable ischemic heart disease, stroke, or NYHA class IV heart failure
* The researchers believe that the patients are compliant insufficiently or not suitable to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
48-week annual recurrence rate (ARR) | 0- 48 weeks
  48-week annual recurrence rate (ARR). ARR is calculated as the total number of relapses for all subjects divided by the total number of years of subjects receiving this treatment

SECONDARY OUTCOMES:
24 weeks confirmed disability progression | 0-24weeks
  Time to 24 weeks confirmed disability progression (24wCDP) (based on EDSS assessment)
12 weeks confirmed disability progression | 0-12weeks
  Time to 12 weeks confirmed disability progression (12wCDP) (based on EDSS assessment)
12 weeks confirmed disability improvement | 0-12weeks
  Time to 12 weeks confirmed disability improvement (12wCDI) (based on EDSS assessment)
Changes in EDSS scores from baseline at weeks 12, 24, 36 and 48 | At 12, 24, 36 and 48 weeks
  Changes in EDSS scores from baseline at weeks 12, 24, 36 and 48; Gadolinium enhanced T1 lesion number in the brain compared with baseline at weeks 12, 24, 36, and 48
Number of new low-signaling T1 lesions in the brain | At 12, 24, 36 and 48 weeks
  Number of new low-signaling T1 lesions in the brain at weeks 12, 24, 36, and 48 compared with baseline
Number of new/new large T2 lesions in the brain | At 12, 24, 36 and 48 weeks
  Number of new/new large T2 lesions in the brain at weeks 12, 24, 36, and 48 compared with baseline
Proportion of patients without recurrence at weeks 0 to 48 | 0- 48 weeks
  Proportion of patients without recurrence at weeks 0 to 48

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital,Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided